CLINICAL TRIAL: NCT05745181
Title: Clinical Study of Anti-CD1a CAR-T in the Treatment of Relapsed Refractory Acute T-lymphoblastic Leukemia/Lymphoblastic Lymphoma
Brief Title: Clinical Study of Anti-CD1a CAR-T in the Treatment of R/R Acute T-lymphoblastic Leukemia/Lymphoblastic Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL479-01
Record Dates: First submitted 2023-02-14; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Acute T-lymphoblastic Leukemia; Acute T-lymphoblastic Lymphoma
Keywords: anti-CD1a CAR-T; relapsed refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T Cell Infusion (Experimental): Peripheral blood mononuclear cells were isolated, amplified and cultured in vitro, pretreated with FC regimen, and Anti-CD1a CAR-T cells were transfused.
  Interventions: Biological: CAR-T Cell Infusion

INTERVENTIONS:
Biological: CAR-T Cell Infusion — Peripheral blood mononuclear cells were isolated, amplified and cultured in vitro, pretreated with FC regimen, and Anti-CD1a CAR-T cells were transfused.

SUMMARY:
To evaluate the efficacy and safety of anti-CD1a CAR-T in the treatment of relapsed refractory acute T-lymphoblastic leukemia/lymphoblastic lymphoma.

DETAILED DESCRIPTION:
Acute T-lymphoblastic leukemia/lymphoblastic lymphoma (T-ALL/LBL) is a highly heterogeneous hematological malignancy usually associated with genetic alterations/mutations in transcription factors that are major regulators of hematopoietic stem/progenitor cell homeostasis and T cell development. 70% of patients develop mass with myeloid invasion and other leukemia symptoms.

CD1a, a transfer membrane glycoprotein, is a cell surface antigen present on cortical T-ALL cells. It is present in 40% of T-ALL cases. Specific expression of this antigen has also been observed in developing cortical thymus cells. It was also slightly expressed in langerhans cells, digital dendritic cells, B lymphocytes and gastrointestinal epithelial cells. CD1a4 was not expressed in CD34+ progenitor cells or T cells during ontogeny. This property of CD1a makes it a suitable target antigen whose targeting minimizes the possibility of non-tumor toxicity.

This study intends to treat r/r CD1a+T-ALL/LBL with CD1a CAR-T to observe its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the informed consent; 2. Male or female patients aged 18-70 years (including 18 and 70 years); 3. The patient was diagnosed with CD1a+ acute T lymphoblastic leukemia/lymphoblastic lymphoma by pathology or flow cytometry, and had no effective treatment options at present, such as chemotherapy or hematopoietic stem cell transplantation after recurrence; Alternatively, the patient voluntarily chooses to administer antiCD1a-CAR T cells as salvage therapy. Inclusion criteria

1. Patients or their legal guardians voluntarily participate and sign the informed consent;
2. Male or female patients aged 18-70 years (including 18 and 70 years);
3. The patient was diagnosed with CD1a+ acute T lymphoblastic leukemia/lymphoblastic lymphoma by pathology or flow cytometry, and had no effective treatment options at present, such as chemotherapy or hematopoietic stem cell transplantation after recurrence; Alternatively, the patient voluntarily chooses to administer antiCD1A-CAR T cells as salvage therapy.
4. The following two categories are included:

(1) CD1a+T lymphoblastic lymphoma (T-LBL); (2) CD1a+ acute T-lymphoblastic leukemia (T-ALL). 5. Subject:

1. There was no remission or residual lesions after treatment, and HSCT (auto/allo-HSCT) was not suitable;
2. Relapse occurred after CR, and HSCT (auto/allo-HSCT) was not suitable;
3. Patients with high risk factors;
4. Relapse or no remission after hematopoietic stem cell transplantation or cellular immunotherapy.

6. Measurable or evaluable lesions; 7. The patient's main tissues and organs function well:

1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤34.2μmol/L;
2. Renal function: creatinine < 220 μmol/L;
3. Lung function: indoor oxygen saturation ≥95%;
4. Cardiac function: left ventricular ejection fraction (LVEF) ≥40%. 8. The patients had not received any anti-cancer treatment such as chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) within the first 4 weeks of enrollment, and their previous treatment-related toxic reactions had recovered to ≤ grade 1 at the time of enrollment (except low toxicity such as hair loss); 9. The patient's peripheral shallow venous blood flow is smooth, which can meet the needs of intravenous infusion; 10. Patients with ECOG score ≤2 and expected survival time ≥3 months. 4. The following two categories are included:

(1) CD1a+T lymphoblastic lymphoma (T-LBL); (2) CD1a+ acute T-lymphoblastic leukemia (T-ALL). 5. Subject:

1. There was no remission or residual lesions after treatment, and HSCT (auto/allo-HSCT) was not suitable;
2. Relapse occurred after CR, and HSCT (auto/allo-HSCT) was not suitable;
3. Patients with high risk factors;
4. Relapse or no remission after hematopoietic stem cell transplantation or cellular immunotherapy.

6. Measurable or evaluable lesions; 7. The patient's main tissues and organs function well:

1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤34.2μmol/L;
2. Renal function: creatinine < 220 μmol/L;
3. Lung function: indoor oxygen saturation ≥95%;
4. Cardiac function: left ventricular ejection fraction (LVEF) ≥40%. 8. The patients had not received any anti-cancer treatment such as chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) within the first 4 weeks of enrollment, and their previous treatment-related toxic reactions had recovered to ≤ grade 1 at the time of enrollment (except low toxicity such as hair loss); 9. The patient's peripheral shallow venous blood flow is smooth, which can meet the needs of intravenous infusion; 10. Patients with ECOG score ≤2 and expected survival time ≥3 months.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or breastfeeding;
2. Men or women who have planned to become pregnant within the last 1 year;
3. The patients were not guaranteed to take effective contraceptive measures (condoms or contraceptives, etc.) within 1 year after enrollment;
4. Patients had uncontrollable infectious diseases within 4 weeks prior to enrollment;
5. Active hepatitis B/C virus;
6. Hiv-infected patients;
7. Suffering from a serious autoimmune disease or immunodeficiency disease;
8. The patient is allergic to antibodies, cytokines and other macromolecular biological drugs;
9. The patient had participated in other clinical trials within 6 weeks prior to enrollment;
10. Systemic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Suffers from mental illness;
12. The patient has substance abuse/addiction;
13. According to the researchers judgment, the patient had other conditions that were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From 2 weeks to 1 year.
  CR+PR
Progression-free survival | From 2 weeks to 1 year.
  The time between treatment and observation of disease progression or death from any cause.
overall survival | From 2 weeks to 1 year.
  The time interval between patient infusion of CAR-T and death from any cause or the end of follow-up.
Event-free survival | From 2 weeks to 1 year.
  The time from the start of CAR-T infusion to the occurrence of any event.

SECONDARY OUTCOMES:
Characterization of the level of CAR T cell expansion in subjects over time | From 2 weeks to 1 year.
  Characterization of the level of CAR T cell expansion in subjects over time.
Duration of CAR T cells in subjects | From 2 weeks to 1 year.
  Duration of CAR T cells in subjects
Characteristics of lymphocyte reduction in subjects | From 2 weeks to 1 year.
  Characteristics of lymphocyte reduction in subjects

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No